CLINICAL TRIAL: NCT04733521
Title: A Phase 1/2, Open-label, Study to Investigate the Safety, Tolerability, and Efficacy of SC-43 Administered in Combination With Cisplatin in Subjects With Advanced or Refractory Non-small Cell Lung Cancer or Biliary Tract Carcinoma
Brief Title: A Phase 1/2 Study of SC-43 in Combination With Cisplatin
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RaND Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-SCR-01
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Advanced Non-small-cell Lung Cancer; Advanced Biliary Tract Cancer
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NSCLC (Experimental)
  Interventions: Drug: SC-43; Drug: Cisplatin
- BTC (Experimental)
  Interventions: Drug: SC-43; Drug: Cisplatin

INTERVENTIONS:
Drug: SC-43 — SC-43 oral, every day of 21-day cycle
Drug: Cisplatin — cisplatin 75mg/m2 on day 1 of 21-day cycle

SUMMARY:
SC-43 is STAT3 inhibitor. Based on the phase I data of SC-43 monotherapy, this is a Phase 1/2, Open-label, Study to Investigate the Safety, Tolerability, and Efficacy of SC-43 Administered in Combination with Cisplatin in Subjects with Advanced or Refractory Non-small Cell Lung Cancer or Biliary Tract Carcinoma

DETAILED DESCRIPTION:
Based on the ongoing Phase 1 study in refractory cancer types, it is deemed adequate to select the starting dose at 50 mg in combination with cisplatin for NSCLC or BTC. The safety monitoring committee (SMC) will review the starting dose of 50 mg data and decide whether it is adequate to escalate the dose to 100, then 150 mg according to Bayesian optimal interval (BOIN) design. Moreover, based on the PK profiles and modelling, the loading dose 100 mg QD for 7 days will keep the minimal efficacy concentration and effectively maintain the p-STAT3 level low enough to translate the anticancer efficacy with clinical efficacy for the study drug SC-43.

The cisplatin efficacy for NSCLC and BTC, the chosen dose and dosing schedules 75 mg/m2 in a 3-week cycle in combination with SC-43 are supported by previous clinical experience of observed efficacy and safety profiles for the indicated study populations.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥ 12 weeks.
* Histologically or cytologically confirmed NSCLC or BTC.
* At least 1 measurable target lesion ≥ 10 mm as measured by MRI or CT according to RECIST v1.1-criteria. Target lesions within the field of prior efficacy irradiation or in the area of local treatment (intervention or ablation therapy) are considered measurable in case of confirmation of progression.
* Optional availability of archival or fresh tumor specimen that is suitable for analysis. Acceptable samples must have been acquired from a surgical operation, using core needle biopsy, or excisional biopsy. Samples that were acquired using fine needle aspiration are not acceptable. Archival samples from the primary or recurrent cancer will have been taken within 5 years prior to screening. formalin fixed, paraffin-embedded tumor
* Presence of all the following clinical laboratory findings at screening:

  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, or hemoglobin ≥ 9 g/dL.
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) unless liver metastasis or BTC in which case ≤ 2.5 × ULN is permitted at the investigator's discretion.
  * For BTC subjects, alkaline phosphatase and gamma-glutamyl transferase ≤ 5 × ULN.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN unless disease (NSCLC with liver metastases or BTC) related, in which case ≤ 5 × ULN is permitted at the investigator's discretion.
  * Creatinine ≤ 1.5 × ULN, or calculated or measured creatinine clearance (CrCl) ≥ 60 mL/min as calculated by the Cockcroft-Gault method, or 24-hour measured urine CrCl ≥ 50 mL/min.
* Eastern Cooperative Oncology Group performance status < 2.
* For subjects with chronic hepatitis B or C
* If a female subject or a female spouse/partner of male subject is of childbearing potential, she must agree to use highly effective contraceptives from signing informed consent to 28 days or 5 half-lives of SC-43, whichever is the longest, after the last dose of study drug administration
* Male subjects should be willing to use a condom (with spermicidal foam/gel/film/cream/suppository) to prevent pregnancy and exposure of a female partner and should refrain from donating sperm or fathering a child from signing informed consent to 90 days after the last dose of study drug administration.
* Able to comprehend and willing to sign an informed consent form (ICF)

Exclusion Criteria:

* Clinically active or untreated central nervous system (CNS) metastases. Subjects with a history of treated CNS metastases that are asymptomatic are eligible.
* Malignancies other than NSCLC or BTC within 5 years prior to study enrollment, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent, or breast ductal carcinoma in situ treated surgically with curative intent).
* Any ≥ grade 2 (according to NCI-CTCAE v 5.0) AE at baseline (other than those previously allowed in the inclusion criteria).
* History of organ or tissue transplantation.
* History of autoimmune disease.
* Any serious acute, chronic infections that require systemic antimicrobial, antifungal, or antiviral therapy at screening, excluding viral hepatitis.
* History of human immunodeficiency virus infection.
* Significant cardiovascular disease, including:

  * Heart disease classified as New York Heart Association class III or IV.
  * Ongoing uncontrolled hypertension.
  * History of congenital long QT syndrome.
  * Ongoing prolonged QT interval corrected for heart rate using Fridericia's method (QTcF) defined as ≥ 470 msec.
  * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation).
  * Subjects with atrial fibrillation, that is well controlled with treatment, can be enrolled.
* Ascertained hypersensitivity to any ingredient of SC-43 or drugs with similar chemical structures, including sorafenib. If there is suspicion that the subject may have an allergy, the subject should be excluded.
* Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily oral SC-43 treatment
* Significant gastrointestinal disorder(s) within 12 weeks prior to screening that would, in the opinion of the investigator, prevent absorption of an orally available agent
* Active bleeding during the last 4 weeks prior to screening or in the investigator's judgment, the existence of high bleeding tendency lesions such as active gastrointestinal ulcers or prominent esophageal or gastric varices.
* Requirement for ongoing immunosuppressive agents (including azathioprine, mycophenolate, cyclophosphamide, chlorambucil, methotrexate, cyclosporine), or systemic steroid with equivalent dosage higher than prednisolone 30 mg/day for more than 14 days.
* Received an investigational agent within 4 weeks prior to screening.
* Had previous anticancer therapy (surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, biological therapy, or hormonal therapy) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the first dose of SC-43

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose(RP2D) of SC-43 | 18 weeks
  to determine a RP2D of SC-43 for each population of non-small cell lung cancer and biliary tract carcinoma subjects
preliminary antitumor activity of SC-43 | 18 weeks
  the preliminary antitumor activity of SC-43 in combination with other anticancer agents as measured by overall response rate (ORR) according to standard criteria (Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1])

SECONDARY OUTCOMES:
incidence of treatment-related adverse events as assessed by NCI-CTCAE v5.0 | 18 weeks
  incidence of treatment-related adverse events in combination with cisplatin in subjects with non-small cell lung cancer and biliary tract carcinoma. All adverse events will be assessed for severity based on NCI-CTCAE version 5.0
Maximum plasma concentration (Cmax) | day 1 of cycle 1, day 1 of cycle 2 (each 21-day cycle)
  PK blood samples will be collected at predefined time intervals, and the maximum plasma concentration will be determined.
Area under the plasma concentration versus time curve (AUC) | day 1 of cycle 1, day 1 of cycle 2 (each 21-day cycle)
  PK blood samples will be collected at predefined time intervals, and the AUC from time 0 to the last time point will be calculated.
Objective response rate (ORR) according to RECIST criteria version 1.1 | 18 weeks
  Objective response rate (ORR) is defined as the proportion of subjects with complete response (CR) or partial response (PR) as best overall response evaluated according to RECIST criteria version 1.1 on MRI or CT results
Disease control rate (DCR) according to RECIST criteria version 1.1 | 18 weeks
  Disease control rate (DCR) is defined as the proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD) as best overall response evaluated according to RECIST criteria version 1.1 on MRI or CT results.
Duration of response(DOR) according to RECIST criteria version 1.1 | 18 weeks
  Duration of response(DOR) is defined as the time between the date of first response and the date of disease progression.
Progression free survival(PFS) according to RECIST criteria version 1.1 | 18 weeks
  progression free survival(PFS) is defined as the time between the date of first dose of SC-43 and the date of progression or death, whichever occurs first
overall survival(OS) according to RECIST criteria version 1.1 | 18 weeks
  overall survival(OS) time is defined as the length of time from the first dose of SC-43 to the date of death, regardless of the cause of death

OTHER OUTCOMES:
phosphorylated signal transducer and activator of transcription 3(p-STAT3) status in peripheral blood mononuclear cells (PBMCs) of subjects | day -14 to -1(prior to dosing), day 1 of cycle 2 and cycle 3, and end of treatment (each 21-day cycle)
  levels of p-STAT3 (with and without cytokine stimulation) before and after dosing

CONTACTS AND LOCATIONS:
Overall Officials: In-Jae Oh, MD, Principal Investigator — Chonnam National University